CLINICAL TRIAL: NCT03978845
Title: Feasibility of Phrenic Nerve Block to Mitigate Self-inflicted Lung Injury in ARF Patients Under Mechanical Ventilation on Spontaneous Breathing
Brief Title: Phrenic Nerve Block to Mitigate Self-inflicted Lung Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE 02029118.2.0000.00.68
Record Dates: First submitted 2019-05-10; First posted 2019-06-07 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2019-05

CONDITIONS: Respiratory Failure; Mechanical Ventilation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Lidocaine; Anesthetics, Local

STUDY DESIGN:
Intervention Model Description: All patients will be submitted to the same procedures. There will be no between-group comparisons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phrenic Nerve Blockade (Experimental): All patients will be submitted to bilateral phrenic nerve block on its cervical portion.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Using an ultrasound and a nerve stimulator, the phrenic nerve will be identified and low-dose lidocaine will be administered perineurally.
  Other Names: Local anesthetic

SUMMARY:
The purpose of this single-centered, proof of concept study is to determine whether it is feasible to perform a phrenic nerve block to reduce diaphragm electrical activity and, therefore, inspiratory effort and if such block reduces self-inflicted lung injury on patients under mechanical ventilation on spontaneous breathing. Ten patients will be monitored with electrical impedance tomography, NAVA catheter, and esophageal balloon. Using a nerve stimulator and an ultrasound, we will identify the phrenic nerve on its cervical portion bilaterally and administer perineural low-dose lidocaine. Diaphragm electrical activity, transpulmonary pressure and data on ventilation distribution will be continuously collected. The study will be over once the patient presents the same diaphragm electrical activity and transpulmonary pressure as before the phrenic nerve block.

DETAILED DESCRIPTION:
The use of protective mechanical ventilation has improved prognosis on patients with Acute Respiratory Failure. The association of neuromuscular blockade in the first 48-72h has additionally contributed to a higher survival rate. Such improvement may be due to the reduction of transpulmonary pressures caused by the patient's inspiratory effort. To achieve appropriate neuromuscular blockade, highes doses of both neuromuscular blocking agents and sedatives are required. Therefore, such a strategy usually causes muscular atrophy, including the diaphragm.

Because of the augmented neural drive of such patients, exacerbated by inflammation and pulmonary edema, the consequent high tidal volume and transpulmonary pressure cannot be reduced by the newest sedatives. In fact, some of these sedatives may even deteriorate ventilatory dyssynchrony. Our intention is to verify a novel approach: whether is possible to reduce the inspiratory effort of patients without the use of systemic neuromuscular blocking agents.

Our objective in this proof of concept study is to determine the feasibility the use of phrenic nerve blockade to decrease transpulmonary pressure and tidal volume, as well as quantify its effects on esophageal pressure, diaphragmatic electrical activity, transpulmonary pressure and ventilation distribution in patients on spontaneous breathing. It is expected that such intervention will reduce diaphragm electrical activity, leading to lower transpulmonary pressure, tidal volume and driving pressures.

All patients will be submitted to the same intervention. Respiratory mechanics, ventilation distribution, diaphragm electrical activity, heart rate, mean arterial pressure and peripheral saturation will be collected throughout the study. Once the patient presents the same diaphragmatic electrical activity and transpulmonary pressure as before the phrenic nerve block, the study will be over.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years-old;
* Under mechanical ventilation on spontaneous breathing, capable of triggering the ventilator with P/F < 300;
* Tidal volume > 10ml/kg with inspiratory pressure of 12 cmH2O OR driving pressure > 15 cm H2O with inspiratory pressure of 12 cmH2O

Exclusion Criteria:

* Use of neuromuscular blocking agents less than 3h;
* Richmond Agitation-Sedation Scale (RASS) > 0;
* Arterial pH < 7.25;
* Hemodynamically unstable or with increasing doses of vasopressors in the last 2h;
* Intracranial hypertension;
* Thoracic or abdominal tubes;
* Any neuromuscular disease;
* Spinal injury;
* Ascitis;
* Thoracic burn injury;
* Tetanus;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Reduction of tidal volume or transpulmonary pressure | 20 minutes
  Tidal volume or transpulmonary pressure measured using EIT, Servo-I and an esophageal balloon

SECONDARY OUTCOMES:
Reduction of the inspiratory effort | 20 minutes - 3 hours
  Diaphragm electrical activity using NAVA
Consequences on mechanical ventilation | 20 minutes - 3 hours
  Tidal volume, pendellfut and asynchronies measured by EIT
Time to complete weaning of the blockade | 30 minutes - 3 hours
  Patients will be monitored until full recover of inspiratory effort or diaphragm electrical activity
Reduction of the inspiratory effort | 20 minutes - 3 hours
  Esophageal pressure using an esophageal catheter

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim E Vieira, MD, PhD, Principal Investigator — University of Sao Paulo School of Medicine; Marcelo BP Amato, MD, PhD, Principal Investigator — University of Sao Paulo School of Medicine
Locations (1):
- Hospital das Clínicas - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No